CLINICAL TRIAL: NCT01303016
Title: Improving Nutrition and Health Outcomes in Intibuca, Honduras
Acronym: MANI II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shoulder to Shoulder (Other)
Collaborators: The Mathile Institute for the Advancement of Human Nutrition (Other)
Responsible Party: Jeff Heck, MD, Executive Director, Shoulder to Shoulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MANI II, Shoulder to Shoulder
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Malnutrition; Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition supplement (Experimental): Receives a month's supply of the nutrition supplement, Chispuditos, in addition to a voucher for 1lb of powdered milk each month and a voucher for 1lb of sugar every other month.
  Interventions: Dietary Supplement: Chispuditos
- Control (No Intervention): Receives a voucher for 1lb of powdered milk each month and a voucher for 1lb of sugar every other month. Participants in the control group will receive the nutrition supplement, Chispuditos, for one year after the study is complete.

INTERVENTIONS:
Dietary Supplement: Chispuditos — Daily dose per child is 1 heaping Tablespoon of Chispuditos (using the appropriate measuring spoon provided to each participant), 1 teaspoon of sugar if desired (using appropriate measuring spoon provided to each participant), mixed with 8 ounces of water or milk. The mixture is stirred over a heat source (fire or stove) until the mixture boils for 8 minutes.
  Arms: Nutrition supplement

SUMMARY:
The purpose of this research study is to better understand how to prevent malnutrition in children under age 5 years in Intibuca, Honduras. A randomized community trial design was used to implement a nutrition program, including a complementary nutrition supplement, educational sessions, and growth and health monitoring integrated into the basic primary care package, to participants living in communities in the intervention group. Participants living in the control group communities will receive the nutrition supplement for one year following the study.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 months and under 5 years at the time enrollment who reside in Concepcion.

Exclusion Criteria:

* Children with congenital anomalies, mental retardation, severe physical handicap, undernutrition caused by medical conditions that contribute to undernutrition such as heart disease, kidney failure, face and throat problems that interfere with swallowing, medical problems interfering with the absorption of food, and chronic diseases such as tuberculosis, etc.
* Plans to move or change place of residence outside the intervention region in the next 2 months.
* Children whose weight for age z score falls below - 3.
* Children whose weight for age z score is above 3.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 639 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Height and weight | Every other month for 12 months
  Participating children are measured and weighed by trained staff every other month during the 12 month intervention.
Hemoglobin | Baseline, month 6, and month 12
  Hemoglobin values are measured using a One STAT Site M meter instrument and recorded to the nearest g/dL at baseline, month 6, and month 12 of the intervention.
Retinol binding protein, transferrin receptor, and C-Reactive Protein | Baseline, month 6, and month 12
  Retinol binding protein, transferrin, and C-Reactive Protein are measured from dried blood spots collected at baseline, month 6, and month 12 of the intervention.

SECONDARY OUTCOMES:
Food insecurity | Baseline, month 6, and month 12
  Assessment teams administer a scored questionnaire at baseline, month 6, and month 12 of the intervention.
Health outcomes | Baseline, month 6, and month 12
  Assessment teams administer a scored questionnaire at baseline, month 6, and month 12 of the intervention.
Acceptability/Sustainability of nutrition supplement | Baseline, month 3, and month 8
  Assessment teams administer a scored questionnaire at baseline, month 3, and month 8 of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Heck, MD, Principal Investigator — Shoulder to Shoulder